CLINICAL TRIAL: NCT06221293
Title: Study of the Relationship Between Intra-abdominal Pressure, Biomarkers of Bacterial Translocation and Intestinal Wall Damage in Multiple Organ Dysfunction Syndrome.
Brief Title: Correlation Between Intra-abdominal Pressure, Biomarkers of Bacterial Translocation and Intestinal Wall Damage
Status: Active, not recruiting | Type: Observational
Sponsor: Karaganda Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: ИРН АР 19677271; ИРН AP19677271 (Other: Karaganda MU)
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Intraabdominal Hypertension; Multi-Organ Disorder; Translocation Syndrome
Keywords: bacterial translocation; presepsin; intraabdominal hypertension; multi-organ disorder; I-FABP; REG3a; Zonulin
MeSH Terms: conditions — Intra-Abdominal Hypertension

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: the first group consists of patients with increased abdominal pressure, signs of multi-organ failure with a fatal outcome
  Interventions: Diagnostic Test: immunoenzyme analysis
- Group 2: the second group consists of patients with increased abdominal pressure, signs of multi-organ failure without death
  Interventions: Diagnostic Test: immunoenzyme analysis

INTERVENTIONS:
Diagnostic Test: immunoenzyme analysis — immunoenzyme analysis with EVOLIS system

SUMMARY:
Main scientific hypotheses of the project:

1. The level of intestinal microflora translocation markers and biomarkers of intestinal wall damage the in the blood serum correlates with the level of intra-abdominal pressure, regardless of the genesis of intra-abdominal hypertension.

2. The critical levels of intestinal microflora translocation markers and biomarkers of the intestinal wall damage can be used for predicting an unfavorable outcome in the multiple organ dysfunction syndrome.

3. The revealed critical level of intra-abdominal pressure is an additional prognostic sign in assessing the course of the multiple organ dysfunction syndrome.

. Project objectives:

1. To evaluate the indicators of biomarkers of translocation of the intestinal microflora and biomarkers of the intestinal wall damage in the systemic circulation during the development and course of the syndrome of multiple organ dysfunction. Based on the obtained critical levels of markers of translocation of the intestinal microflora and markers of the intestinal wall damage, it will be possible to predict adverse outcomes in patients with multiple organ dysfunction syndrome.
2. To identify differences in the level of markers of bacterial translocation of the intestinal microflora and the level of markers of the intestinal wall damage in patients with intra-abdominal hypertension. In patients with multiple organ dysfunction syndrome, the levels of biomarkers of bacterial translocation of the intestinal microflora and biomarkers of intestinal wall damage in the blood serum correlate with intra-abdominal pressure indicators, regardless of the etiology of intra-abdominal hypertension.
3. Assess the impact of the level of intra-abdominal pressure on the development and course of the syndrome of multiple organ dysfunction. To assess the course of the syndrome of multiple organ dysfunction, an additional prognostic marker is the determination of the critical level of intra-abdominal pressure.
4. Determine the critical levels of biomarkers of intestinal microflora translocation and biomarkers of intestinal wall damage to predict the outcome of diseases accompanied by the development of multiple organ dysfunction syndrome. The obtained critical levels of biomarkers of translocation of the intestinal microflora and biomarkers of the intestinal wall damage will be significant indicators in the syndrome of multiple organ dysfunction for predicting an unfavorable outcome.

DETAILED DESCRIPTION:
The aim of the project is to evaluate the impact of intra-abdominal hypertension, biomarkers of bacterial translocation and biomarkers of intestinal wall damage on the course and outcomes of the disease in patients with multiple organ dysfunction.

Today the intestinal microflora translocation is considered as one of the key mechanism of an enhanced systemic inflammatory response that leads to multiple organ dysfunction. In the intensive care unit, in patients in serious condition changes in various body systems develop, including the immune system reacts with the production of endogenous pro-inflammatory mediators, and due to microcirculation disorders, ischemia and hypoxia of the intestinal wall, aggravated by an increase in intra-abdominal pressure, its permeability increases, its barrier function is impaired. As a result, bacteria and/or their endotoxins penetrate the damaged intestinal barrier and further enhance the immune response, which becomes systemic and ultimately leads to multiple organ dysfunction. When the described processes occur, the assessment of splanchnic blood flow becomes especially relevant.

sCD14-ST (presepsin) and LBP (lipopolysaccharide-binding protein) are being studied as biomarkers of bacterial translocation, and I-FABP (Intestinal fatty-acid binding protein), REG3α (regenerating islet-derived protein-3α) and Zonulin (zonulin) are being studied as biomarkers of intestinal wall injury.

The interaction of the macrophage membrane protein CD14 with peptidoglycans of gram-positive and lipopolysaccharides of the walls of gram-negative bacteria leads to the production of sCD14-ST. Presepsin is a biomarker for the early phase of sepsis and a predictor of outcome in septic patients.

LBP increases the sensitization of receptors of cells of the immune system: macrophages, monocytes, neutrophils to bacterial lipopolysaccharide, which leads to the activation of the immune response by releasing pro-inflammatory mediators. LBP appears to be an effective biomarker for bacterial translocation and the development of septic complications.

I-FABP is a protein that is located on the villi of mature enterocytes. An increase in the level of I-FABP in the blood serum is associated with a violation of the permeability of the intestinal wall, which has been proven in a number of studies.

Paneth cells secrete the antimicrobial protein REG3α into the intestine, and in case of the intestinal wall damage, it moves into the bloodstream. This protein is a reliable biomarker of intestinal wall damage.

Zonulin is a protein that playing a significant role in intestinal wall permeability. It opens the intracellular tight junctions between the cells of the duodenum and small intestine, which leads to an increase in the permeability of the intestinal wall. Therefore, serum zonulin is a marker of dysfunction and increased permeability of the intestinal barrier.

In the databases of publications (Scopus, Web of Science) there were no articles on the study of the relationship between the level of biomarkers of intestinal translocation, the level of biomarkers of the intestinal wall damage and the level of intra-abdominal pressure in patients with multiple organ dysfunction syndrome. This study will allow a more in-depth study of the pathogenesis of intestinal microflora translocation in patients with multiple organ dysfunction syndrome, and will also allow using the results obtained to predict the course of this condition.

Detection of blood serum biomarkers sCD14-ST, LBP, I-FABP, REG3α and Zonulin will be performed by enzyme immunoassay. The level of intra-abdominal pressure will be measured by the method of tonometry in the bladder through a urethral catheter using a portable invasive low pressure meter (IIND - 500/75) by Triton-Electronics LLC.

The expected scientific results of studying the relationship between intra-abdominal pressure, the phenomenon of translocation of intestinal microflora into the systemic circulation with the pathogenesis and dynamics of the development of multiple organ dysfunction syndrome will have an impact on the further improvement of the treatment tactics of this pathology. Innovative methods for diagnosing the phenomenon of intestinal microflora translocation will have a positive effect on the development of laboratory diagnostics and science in Kazakhstan.

Revealing of relationships between intestinal microflora translocation biomarkers, biomarkers of the intestinal wall damage and changes in intra-abdominal pressure will allow a more in-depth study of the pathogenetic mechanisms in the development and course of the multiple organ dysfunction syndrome, depending on its genesis, which will allow using the results obtained to predict the outcomes of this syndrome.

2.2. The aim of the project is to evaluate the impact of intra-abdominal hypertension, biomarkers of bacterial translocation, and biomarkers of the intestinal wall damage on the course and outcomes of the disease in patients with multiple organ dysfunction.

2.3. Project objectives:

1. To evaluate the indicators of biomarkers of translocation of the intestinal microflora and biomarkers of the intestinal wall damage in the systemic circulation during the development and course of the syndrome of multiple organ dysfunction. Based on the obtained critical levels of markers of translocation of the intestinal microflora and markers of the intestinal wall damage, it will be possible to predict adverse outcomes in patients with multiple organ dysfunction syndrome.
2. To identify differences in the level of markers of bacterial translocation of the intestinal microflora and the level of markers of the intestinal wall damage in patients with intra-abdominal hypertension. In patients with multiple organ dysfunction syndrome, the levels of biomarkers of bacterial translocation of the intestinal microflora and biomarkers of intestinal wall damage in the blood serum correlate with intra-abdominal pressure indicators, regardless of the etiology of intra-abdominal hypertension.
3. Assess the impact of the level of intra-abdominal pressure on the development and course of the syndrome of multiple organ dysfunction. To assess the course of the syndrome of multiple organ dysfunction, an additional prognostic marker is the determination of the critical level of intra-abdominal pressure.
4. Determine the critical levels of biomarkers of intestinal microflora translocation and biomarkers of intestinal wall damage to predict the outcome of diseases accompanied by the development of multiple organ dysfunction syndrome. The obtained critical levels of biomarkers of translocation of the intestinal microflora and biomarkers of the intestinal wall damage will be significant indicators in the syndrome of multiple organ dysfunction for predicting an unfavorable outcome.

3. Scientific novelty and significance of the project Multiple Organ Dysfunction Syndrome (MODS) is a potentially reversible physiological disorder involving two or more organ systems not involved in the process resulting in intensive care unit (ICU) hospitalization. MODS results in longer ICU stays and, in severe cases, leads to high mortality (27%-100%).

In this scientific project, it is planned to study the levels of biomarkers of bacterial translocation (sCD14-ST, LBP) levels of biomarkers of intestinal wall damage (I-FABP, REG3α and Zonulin) and intra-abdominal pressure in patients with multiple organ dysfunction syndrome.

The interaction of the macrophage membrane protein CD14 with peptidoglycans of gram-positive and lipopolysaccharides of the walls of gram-negative bacteria leads to the production of sCD14-ST . Presepsin is a biomarker for the early phase of sepsis and a predictor of outcome in septic patients.

LBP increases the sensitization of receptors of cells of the immune system: macrophages, monocytes, neutrophils to bacterial lipopolysaccharide, which leads to the activation of the immune response by releasing pro-inflammatory mediators. LBP appears to be an effective biomarker for bacterial translocation and the development of septic complications.

I-FABP is a protein that is located on the villi of mature enterocytes. An increase in the level of I-FABP in the blood serum is associated with a violation of the permeability of the intestinal wall, which has been proven in a number of studies.

Paneth cells secrete the antimicrobial protein REG3α into the intestine, and in case of the intestinal wall damage, it moves into the bloodstream. This protein is a reliable biomarker of intestinal wall damage and bacterial translocation.

Zonulin first described like it is a protein that playing a significant role in intestinal wall permeability. It opens the intracellular tight junctions between the cells of the duodenum and small intestine, which leads to an increase in the permeability of the intestinal wall. Therefore, serum zonulin is a marker of dysfunction and increased permeability of the intestinal barrier.

3. Research methods The type of research being conducted is fundamental research. The design of the study complies with the principles of the Declaration of Helsinki of the World Medical Association and was approved by the Local Commission on Bioethics of the NJSC KMU. Clinical bases in Karaganda, where biological material will be taken: Multidisciplinary Hospital No. 1, Regional Clinical Hospital, Clinic of Medical University. Laboratory research will be carried out on the basis of the Research Laboratory of the Institute of Life Sciences of the NJSC KMU.

Main scientific hypotheses of the project:

1. The level of intestinal microflora translocation markers and biomarkers of intestinal wall damage the in the blood serum correlates with the level of intra-abdominal pressure, regardless of the genesis of intra-abdominal hypertension.
2. The critical levels of intestinal microflora translocation markers and biomarkers of the intestinal wall damage can be used for predicting an unfavorable outcome in the multiple organ dysfunction syndrome.
3. The revealed critical level of intra-abdominal pressure is an additional prognostic sign in assessing the course of the multiple organ dysfunction syndrome.

Research material. It is planned to study bacterial translocation biomarkers (sCD14-ST, LBP), biomarkers of intestinal wall damage (I-FABP, REG3α and Zonulin) in blood serum and measure intra-abdominal pressure in 180 patients with multiple organ dysfunction syndrome.

Measurement of intra-abdominal pressure will be carried out in patients with multiple organ dysfunction syndrome through a urethral catheter using a portable electronic device "ILPM - 500/75" (invasive low-pressure meter) manufactured by LLC "Triton - ElectronicS", Yekaterinburg, RF.

Technique for measuring intra-abdominal pressure: 50 ml of warm sterile isotonic sodium chloride solution is injected into the previously emptied bladder through a Foley catheter with an inflated balloon using a syringe without a needle. The urethral catheter is attached to the measuring device. With the valve of the urethral catheter closed, a zero value is set, after which the valve of the catheter is opened and the intra-abdominal pressure is recorded according to the indication on the display of the device

Risks and their solutions:

1. With an increase in prices for the necessary reagents and materials due to the constant change in the exchange rate, most of the purchase will be carried out in the 1st year of the project implementation. Reducing the number of studies conducted while maintaining statistical significance without significant losses for the project.
2. When changing the place and dates of congresses and conferences with a change in travel costs, there will be changes in the number of business travelers.

ELIGIBILITY:
Inclusion Criteria:

* registered multiple organ dysfunction syndrome of various genesis
* over 18 years of age.

Exclusion Criteria:

* age under 18
* pregnancy
* HIV infection

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age with multi-organ dysfunction syndrome and increased intra-abdominal pressure
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2025-12-27 (Estimated)

PRIMARY OUTCOMES:
Detection of biomarkers of translocation | 3-10 days
  To evaluate the indicators of biomarkers of translocation of the intestinal microflora and biomarkers of the intestinal wall damage in the systemic circulation during the development and course of the syndrome of multiple organ dysfunction. Based on the obtained critical levels of markers of translocation of the intestinal microflora and markers of the intestinal wall damage, it will be possible to predict adverse outcomes in patients with multiple organ dysfunction syndrome.

SECONDARY OUTCOMES:
The differences between level of bacterial translocation and level of markers of the intestinal wall damage with intraabdominal hypertension | 3-10 days
  To identify differences in the level of markers of bacterial translocation of the intestinal microflora and the level of markers of the intestinal wall damage in patients with intra-abdominal hypertension. In patients with multiple organ dysfunction syndrome, the levels of biomarkers of bacterial translocation of the intestinal microflora and biomarkers of intestinal wall damage in the blood serum correlate with intra-abdominal pressure indicators, regardless of the etiology of intra-abdominal hypertension.

OTHER OUTCOMES:
Correlation between the level of intraabdominal hypertension and progression of multi-organ dysfunction | 3-10 days
  Assess the impact of the level of intra-abdominal pressure on the development and course of the syndrome of multiple organ dysfunction. To assess the course of the syndrome of multiple organ dysfunction, an additional prognostic marker is the determination of the critical level of intra-abdominal pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Alina Ogizbaeva, dr, Principal Investigator — young scientist, phD; Kairat Shakeyev, dr, Principal Investigator — head of the surgical service of the CSE "Multidisciplinary Hospital No. 3 of Karaganda; Dmitry Matyushko, dr, Principal Investigator — PhD, Associate Professor of the Department of Surgical Diseases; Miras Mugazov, dr, Principal Investigator — PhD, Associate Professor of the Department of Emergency Medical Care; Dana Amanova, dr, Study Chair — PhD, young scientist, co-investigator; Zhibek Zhumadilova, Study Chair — young scientist, co-investigator; Shynggys Nuraly, Study Chair — young scientist, co-investigator; Sofiko Assamidanova, Study Chair — young scientist, co-investigator; Yermek Turgunov, dr, Study Director — professor
Locations (5):
- Kazakhstan (5):
  - Karaganda Medical University, Karaganda
  - Clinic of the Medical University of Karaganda, Karaganda
  - Multidisciplinary hospital No. 1, Karaganda
  - Multidisciplinary Hospital No. 3, Karaganda
  - Regional Clinic Hospital, Karaganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Turgunov Y, Ogizbayeva A, Akhmaltdinova L, Shakeyev K. Lipopolysaccharide-binding protein as a risk factor for development of infectious and inflammatory postsurgical complications in colorectal cancer paients. Contemp Oncol (Pozn). 2021;25(3):198-203. doi: 10.5114/wo.2021.110051. Epub 2021 Oct 14. PMID 34729040
- [Result] Shakeyev K, Turgunov Y, Ogizbayeva A, Avdiyenko O, Mugazov M, Grigolashvili S, Azizov I. Presepsin (soluble CD14 subtype) as a risk factor for the development of infectious and inflammatory complications in operated colorectal cancer patients. Ann Coloproctol. 2022 Dec;38(6):442-448. doi: 10.3393/ac.2022.00115.0016. Epub 2022 Apr 4. PMID 35368178
- [Result] Amanova DY, Lavrinenko AV, Kaliyeva DK, Matyushko DN, Ivachyov PA, Turgunov YM. Comparative Evaluation of Translocation of GFP Producing Escherichia coli Strains in Acute Intestinal Obstruction. Bull Exp Biol Med. 2019 Sep;167(5):660-662. doi: 10.1007/s10517-019-04593-y. Epub 2019 Oct 17. PMID 31625067
- [Result] Ivachyov P, Amanova D, Akhmaltdinova L, Koishibayev Z, Turgunov E. [COMPARISON OF DYNAMICS OF LEVEL OF PROCALCITONIN, LIPOPOLYSACCHARIDE BINDING PROTEIN AND INTERLEUKIN-6 IN BLOOD SERUM OF EXPERIMENTAL ANIMALS AT STRANGULATED AND OBTURATIVE INTESTINAL OBSTRUCTION]. Georgian Med News. 2020 Jun;(303):173-177. Russian. PMID 32841201
- See also: Annals of Coloproctology 2022;38(6):442-448 — http://www.coloproctol.org/journal/view.php?number=1925
- See also: J CLIN MED KAZ, Volume 18, Issue 3, pp. 8-13. — http://www.clinmedkaz.org/article/bacterial-translocation-in-colorectal-cancer-patients-10926
- See also: J CLIN MED KAZ, Volume 19, Issue 2, pp. 38-42. — http://www.clinmedkaz.org/article/the-16s-ribosomal-ribonucleic-acid-microorganisms-detection-in-mesenteric-lymph-nodes-by-a-11937